CLINICAL TRIAL: NCT03587259
Title: Innovation in Mammography: Tomosynthesis Pathways
Acronym: IMPETO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Prevention and Research Institute, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: F16J16000620002
Record Dates: First submitted 2018-06-27; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
Keywords: breast cancer screening; tomosynthesis; digital mammography
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2D mammography (Active Comparator): 45-46 years old women are invited to attend the usual screening examination (2D mammography). The next year they will be invited to make a 2D mammography, according to screening protocol.
  Interventions: Diagnostic Test: 2D mammography
- Tomosynthesis (Experimental): 45-46 years old women are invited to attend the Digital Breast Tomosynthesis (DBT) in adjunct to synthetic mammograms (sDM). The next year they will be invited to make a 2D mammography, according to screening protocol.
  Interventions: Diagnostic Test: Tomosynthesis

INTERVENTIONS:
Diagnostic Test: Tomosynthesis — DBT is a x-ray examination that allows to visualize the breast on 3 planes (3D) and therefore to help to see lesions hardly visible to mammography due to the overlap of glandular tissue.
  Other Names: Digital Breast Tomosynthesis (DBT)
  Arms: Tomosynthesis
Diagnostic Test: 2D mammography — 2D mammography is a X-ray examinations used to detect breast cancer in the screening programme.
  Arms: 2D mammography

SUMMARY:
The study aims at evaluating the introduction of tomosynthesis in mammography screening, analyzing the benefits, disadvantages and feasibility in current clinical practice.

It involves women aged 45-46 that will be divided, by drawing lots, into two groups: one group will do the 2D digital mammography (control group), while the other group (intervention group) will do tomosynthesis. In the intervention group the 2D two-dimensional mammography will be reconstructed starting from tomosynthesis without exposing women to other radiation.

DETAILED DESCRIPTION:
The IMPETO trial is a population-based, multicentre, randomised trial aimed at evaluating the clinical accuracy of Digital Breast Tomosynthesis (DBT) in adjunct to synthetic mammograms (sDM) compared to standard two-dimensional digital mammography alone (2D) in a screening programme.

45-46 year-old women resident in the screening centre catchment area of Florence and South-Est Local Health Unit are invited to attend for mammography screening and asked for informed consent to be included in the study. Women are then randomly allocated either to an usual care group (2D mammography) or to the intervention group. In the intervention group, DBT combined with sDM is proposed in order to reduce radiation exposure. The next year women of both groups will be invited to attend the usual screening examination (2D mammography). The enrolment will last 12-18 months; the whole study 36 months. The estimated sample size is 6000 women, 3000 per arm. Data will be pooled with the trial "Screening for Breast Cancer With Digital Breast Tomosynthesis", ClinicalTrials.gov Identifier: NCT02698202.

ELIGIBILITY:
Inclusion Criteria:

* 45-46 years old women resident in the screening area

Exclusion Criteria:

* previous breast cancer
* written refusal to participate in the screening programme
* pregnancy, breastfeeding
* presence of prostheses;
* ongoing chemotherapy;
* impossibility to submit the informed consent for linguistic problems or for inability of women to provide informed consent;
* verified presence of BRCA1 - BRCA2 (Breast Related Cancer Antigens 1 - Breast Related Cancer Antigens 2) genetic mutation or involvement in surveillance path for heredo-familial tumor;
* previous known tomosynthesis.

Ages: 45 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6000 (Estimated)
Dates: Start 2018-09-03 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
the cumulative incidence of advanced screen-detected cancers (T2 +) and the cumulative incidence of advanced interval cancers (T2 +) | three years
  number of T2+ screen-detected cancers divided by all screened women at subsequent round of screening and number of T2+ interval cancers divided by all screened women at subsequent round of screening.

SECONDARY OUTCOMES:
recall rate | two years
  number of women recalled to perform 2nd level assessments) for invasive tests and for non-invasive examinations in the two arms divided by the number of screened women
detection rate | two years
  number of breast cancer cases (invasive and in situ forms) divided by the number of screened women (per 1,000)
benign biopsies rate | two years
  number of benign biopsies divided by the total number of biopsies
cost analysis | two years
  an activity based cost analysis will be performed in order to obtain the real costs of DBT screening pathway.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Mantellini, MDr, Principal Investigator — Oncological Network, Prevention and Research Institute
Locations (2):
- Italy (2):
  - South-Est Local Health Unit, Arezzo
  - Oncological Network, Prevention and Research Institute, Florence

REFERENCES:
- [Background] Ciatto S, Houssami N, Bernardi D, Caumo F, Pellegrini M, Brunelli S, Tuttobene P, Bricolo P, Fanto C, Valentini M, Montemezzi S, Macaskill P. Integration of 3D digital mammography with tomosynthesis for population breast-cancer screening (STORM): a prospective comparison study. Lancet Oncol. 2013 Jun;14(7):583-9. doi: 10.1016/S1470-2045(13)70134-7. Epub 2013 Apr 25. PMID 23623721
- [Background] Skaane P, Bandos AI, Gullien R, Eben EB, Ekseth U, Haakenaasen U, Izadi M, Jebsen IN, Jahr G, Krager M, Niklason LT, Hofvind S, Gur D. Comparison of digital mammography alone and digital mammography plus tomosynthesis in a population-based screening program. Radiology. 2013 Apr;267(1):47-56. doi: 10.1148/radiol.12121373. Epub 2013 Jan 7. PMID 23297332
- [Background] Gilbert FJ, Tucker L, Gillan MG, Willsher P, Cooke J, Duncan KA, Michell MJ, Dobson HM, Lim YY, Purushothaman H, Strudley C, Astley SM, Morrish O, Young KC, Duffy SW. The TOMMY trial: a comparison of TOMosynthesis with digital MammographY in the UK NHS Breast Screening Programme--a multicentre retrospective reading study comparing the diagnostic performance of digital breast tomosynthesis and digital mammography with digital mammography alone. Health Technol Assess. 2015 Jan;19(4):i-xxv, 1-136. doi: 10.3310/hta19040. PMID 25599513
- [Background] Skaane P, Bandos AI, Eben EB, Jebsen IN, Krager M, Haakenaasen U, Ekseth U, Izadi M, Hofvind S, Gullien R. Two-view digital breast tomosynthesis screening with synthetically reconstructed projection images: comparison with digital breast tomosynthesis with full-field digital mammographic images. Radiology. 2014 Jun;271(3):655-63. doi: 10.1148/radiol.13131391. Epub 2014 Jan 24. PMID 24484063
- [Background] Paci E, Mantellini P, Giorgi Rossi P, Falini P, Puliti D; TBST Working Group. [Tailored Breast Screening Trial (TBST)]. Epidemiol Prev. 2013 Jul-Oct;37(4-5):317-27. Italian. PMID 24293498
- [Background] McDonald ES, McCarthy AM, Akhtar AL, Synnestvedt MB, Schnall M, Conant EF. Baseline Screening Mammography: Performance of Full-Field Digital Mammography Versus Digital Breast Tomosynthesis. AJR Am J Roentgenol. 2015 Nov;205(5):1143-8. doi: 10.2214/AJR.15.14406. PMID 26496565
- [Background] Bernardi D, Ciatto S, Pellegrini M, Anesi V, Burlon S, Cauli E, Depaoli M, Larentis L, Malesani V, Targa L, Baldo P, Houssami N. Application of breast tomosynthesis in screening: incremental effect on mammography acquisition and reading time. Br J Radiol. 2012 Dec;85(1020):e1174-8. doi: 10.1259/bjr/19385909. PMID 23175484
- [Background] Bernardi D, Belli P, Benelli E, Brancato B, Bucchi L, Calabrese M, Carbonaro LA, Caumo F, Cavallo-Marincola B, Clauser P, Fedato C, Frigerio A, Galli V, Giordano L, Giorgi Rossi P, Golinelli P, Morrone D, Mariscotti G, Martincich L, Montemezzi S, Naldoni C, Paduos A, Panizza P, Pediconi F, Querci F, Rizzo A, Saguatti G, Tagliafico A, Trimboli RM, Zappa M, Zuiani C, Sardanelli F. Digital breast tomosynthesis (DBT): recommendations from the Italian College of Breast Radiologists (ICBR) by the Italian Society of Medical Radiology (SIRM) and the Italian Group for Mammography Screening (GISMa). Radiol Med. 2017 Oct;122(10):723-730. doi: 10.1007/s11547-017-0769-z. Epub 2017 May 25. PMID 28540564
- [Background] Lang K, Andersson I, Rosso A, Tingberg A, Timberg P, Zackrisson S. Performance of one-view breast tomosynthesis as a stand-alone breast cancer screening modality: results from the Malmo Breast Tomosynthesis Screening Trial, a population-based study. Eur Radiol. 2016 Jan;26(1):184-90. doi: 10.1007/s00330-015-3803-3. Epub 2015 May 1. PMID 25929946
- [Background] Lang K, Nergarden M, Andersson I, Rosso A, Zackrisson S. False positives in breast cancer screening with one-view breast tomosynthesis: An analysis of findings leading to recall, work-up and biopsy rates in the Malmo Breast Tomosynthesis Screening Trial. Eur Radiol. 2016 Nov;26(11):3899-3907. doi: 10.1007/s00330-016-4265-y. Epub 2016 Mar 4. PMID 26943342